CLINICAL TRIAL: NCT04952415
Title: the Prognosis of Fetoscopy Treatment of Twin Transfusion Syndrome in Shengjing Hospital
Brief Title: the Prognosis of Fetoscopy Treatment of Twin Transfusion Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caixia Liu, Director of the second obstetrical department, Shengjing Hospital
Other Study IDs: PFTTTTS
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Twin Diseases
Keywords: TTTS
MeSH Terms: conditions — Diseases in Twins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fetal medicine in China is still a new, young discipline, and the development is very rapid. After nearly 10 years of development, the clinical diagnosis and treatment guidelines of some complicated twin diseases has been established. Among them, twin-to-twin-transfusion syndrome (TTTS) is serious disease in twin pregnancy, and the factors affecting prognosis after fetoscopic laser surgery are part of the study. Through this study, the investigators expect to achieve better prediction indicators of the prognosis of TTTS.

DETAILED DESCRIPTION:
A better guideline for twin-to-twin-transfusion syndrome are anticipated to be established in China. Fetoscopic laser surgery is applied to treat TTTS. After surgery, better prediction indicators of the prognosis of TTTS are needed.

ELIGIBILITY:
Inclusion Criteria:

TTTS after fetoscopic laser surgery.

Exclusion Criteria:

Pregnant women who refuse to take part in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: TTTS after fetoscopic laser surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Weight in kilogram of neonate | At birth of neonate
  Including twin pregnancy of TTTS after fetoscopic laser surgery measured by nurses

SECONDARY OUTCOMES:
Neurodevelopment at early childhood | At age of 1 year old
  Including adaptive, gross motor, fine motor, language, and social function; assessed using Gesell Developmental Schedules.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No